CLINICAL TRIAL: NCT05338086
Title: A Randomised, Double-blind, Parallel, Multinational Study to Compare the Efficacy, Pharmacokinetics, Pharmacodynamics, Safety and Immunogenicity of MB09 (Proposed Denosumab Biosimilar) vs. Prolia® (EU-sourced) in Postmenopausal Osteoporosis
Brief Title: A Study to Compare Efficacy, PK, PD, Safety and IMM of MB09 to Prolia® [EU-sourced] in Postmenopausal Osteoporosis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB09-C-01-19
Record Dates: First submitted 2022-04-08; First posted 2022-04-20 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-12

CONDITIONS: Postmenopausal Women With Osteoporosis
MeSH Terms: interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MB09-MB09 (Experimental): Subjects randomised into MB09-MB09 group were administered MB09 (60 mg in 1 mL) SC injection every 6 months.
  Interventions: Drug: MB09 (denosumab biosimilar); Dietary Supplement: Elemental Calcium; Dietary Supplement: Vitamin D
- Prolia-MB09 (Active Comparator): Subjects randomised into Prolia- MB09 group were administered Prolia® (60 mg in 1 mL) SC injection every 6 months.
  Interventions: Drug: MB09 (denosumab biosimilar); Drug: EU-Prolia; Dietary Supplement: Elemental Calcium; Dietary Supplement: Vitamin D
- Prolia-Prolia (Active Comparator): Subjects randomised into Prolia-Prolia group were administered Prolia® (60 mg in 1 mL) SC injection every 6 months.
  Interventions: Drug: EU-Prolia; Dietary Supplement: Elemental Calcium; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: MB09 (denosumab biosimilar) — Pre-filled syringe (PFS) 60 mg/mL solution, administered as subcutaneous injection
  Arms: MB09-MB09; Prolia-MB09
Drug: EU-Prolia — PFS 60 mg/mL solution, administered as subcutaneous injection
  Arms: Prolia-MB09; Prolia-Prolia
Dietary Supplement: Elemental Calcium — at least 1000 mg daily
Dietary Supplement: Vitamin D — at least 400 IU daily

SUMMARY:
This was a randomized, double-blind, parallel, multicenter, multinational study to compare the efficacy, pharmacokinetics, pharmacodynamics, safety and immunogenicity of MB09 versus Prolia® in postmenopausal women with osteoporosis

DETAILED DESCRIPTION:
The study was planning to randomise approximately 528 postmenopausal women with osteoporosis aged ≥55 and ≤80 years old with a Bone Mineral Density (BMD) consistent with T-score of ≤ -2.5 and ≥ -4 at the lumbar spine or total hip as measured by DXA during the Screening Period. Screening evaluations were to be completed within 28 days prior to randomisation.

On Day 1, 528 eligible postmenopausal women with osteoporosis were to be randomised in a 2:1:1 ratio to receive MB09-MB09 (Arm 1), Prolia-MB09 (Arm 2), or Prolia-Prolia (Arm 3) using an Interactive Response Sys-tem (IRT).

During the Main Treatment Period, subjects received one subcutaneous injection (60 mg/mL) of study drug on Day 1 and at Month 6. At Month 12, after all efficacy and safety assessments have been performed, the subject were to be enter the Transition/Safety Follow Up Period and were to receive the third dose of study drug. Subjects assigned to the MB09 MB09 arm (Arm 1) received MB09 on Day 1, at Month 6 and at Month 12. Subjects assigned to the Prolia MB09 arm (Arm 2) received EU-Prolia on Day 1 and at Month 6, and MB09 at Month 12. Subjects assigned to the Prolia-Prolia arm (Arm 3) received EU-Prolia on Day 1, at Month 6, and at Month 12. All subjects were to be followed up to Transition Period Month 6.

All subjects received daily supplementation of calcium and vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, diagnosed with osteoporosis.
* Aged ≥ 55 and ≤ 80 years at screening.
* Body weight ≥ 50 kg and ≤ 99.9 kg, and a body mass index of ≤30 kg/m2 at screening.
* Absolute bone mineral density consistent with T-score ≤ -2.5 and ≥ -4.0 at the lumbar spine or total hip as measured by Dual-energy X-ray Absorptiometry (DXA).
* At least two intact, nonfractured vertebrae in the L1-L4 region and at least one hip joint evaluable by DXA.
* Adequate organ function.

Exclusion Criteria:

* Previous exposure to denosumab (Prolia®, Xgeva®, or denosumab biosimilar) or other monoclonal antibody.
* History and/or presence of one severe or more than two moderate vertebral fractures or hip fracture.
* Recent long bone fracture (within 6 months).
* History and/or presence of bone metastases, bone disease or other metabolic disease.
* Intravenous bisphosphonate administered within 5 years of screening.
* Oral bisphosphonates ≥12 months cumulative use prior to screening. If used <12 months cumulatively and the last dose was ≥12 months before screening, the subject could be enrolled.
* Ongoing use of any osteoporosis treatment or use of prohibited treatment.
* Other bone active drugs.
* History and/or current hypoparathyroidism or hyperparathyroidism, hypocalcemia or hypercalcemia.
* Other Inclusion/exclusion criteria may apply.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 558 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (64):
- Bulgaria (12):
  - AES - DRS - Medical Center Synexus Sofia EOOD, Sofia, Sofia-Grad
  - Medical Center Medconsult Pleven OOD, Pleven
  - Medical Center Artmed OOD, Plovdiv
  - Multiprofile Hospital for Active Treatment Plovdiv, Plovdiv
  - Outpatient Clinic for Specialized Medical Help - Medical Center Kuchuk Paris "OOD", Plovdiv
  - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia
  - Diagnostic- Consultative Center Convex EOOD, Sofia
  - Medical Center Excelsior OOD - PPDS, Sofia
  - Medical Center Hera EOOD, Sofia
  - Specialized outpatient medical facility - Rheumatology Centre St. Irina EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment - Prof. Dr. Stoyan Kirkovich AD, Stara Zagora
  - New Medical Center EOOD, Vratsa
- Estonia (7):
  - Center For Clinical And Basic Research, Tallinn, Harju
  - East Tallinn Central Hospital, Tallinn, Harju
  - North Estonia Medical Centre Foundation, Tallinn, Harju
  - KLV Arstikabinet, Pärnu, Pärnu Maakon
  - Clinical Research Centre Ltd, Tartu, Tartu
  - MediTrials OÜ, Tartu, Tartu
  - Tartu University Hospital, Tartu, Tartu
- Georgia (3):
  - National Institute of Endocrinology, Tbilisi
  - Tbilisi Heart and Vascular Clinic Ltd, Tbilisi
  - Tbilisi Heart Center Ltd., Tbilisi
- Hungary (11):
  - Bekes Megyei Kozponti Korhaz, Békéscsaba, Bekes County
  - AES - DRS - Synexus Gyula - Magyarország Egészségügyi Szolgáltató Kft, Gyula, Bekes County
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Szentes, Csongrád megye
  - AES - DRS - Synexus Debrecen Magyarország Egészségügyi Szolgáltató Kft, Debrecen, Hajdú-Bihar
  - MÁV Kórház és Rendelointézet Szolnok, Szolnok, Jász-Nagykun-Szolnok
  - Pest Megyei Flór Ferenc Kórház, Kistarcsa, Pest County
  - AES - DRS - Synexus Zalaegerszeg Magyarország Egészségügyi Kft, Zalaegerszeg, Zala County
  - AES - DRS - Synexus Budapest - Magyarország Egészségügyi Szolgáltató Kft, Budapest
  - QUALICLINIC Kft, Budapest
  - Óbudai Egészségügyi Centrum Kft, Budapest
  - Vital Medical Center, Veszprém
- Latvia (5):
  - Private Practice of Laila Atike, Liepāja, Liepājas Rajon
  - Outpatient Clinic Veselibas Centrs 4, Riga, Riga Rajon
  - Outpatient Clinic Adoria, Riga, Rigas Rajons
  - Sigulda Hospital, Outpatient Clinic, Sigulda, Siguldas Pilsēta
  - RSU Ambulance, Riga
- Mexico (5):
  - Centro de Estudios de Investigacion Basica Y Clinica SC, Guadalajara, Jalisco
  - Hospital Angeles Lindavista (Consultorio de Reumatologia), Mexico City, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio González, Monterrey, Nuevo León
  - Centro Integral Medico SJR S.C, Querétaro
  - Hospital Central Dr Ignacio Morones Prieto, San Luis Potosí City
- Poland (17):
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Globe Badania Kliniczne Spólka z o.o., Kłodzko, Lower Silesian Voivodeship
  - Lubelskie Centrum Diagnostyczne (Lotników Polskich), Świdnik, Lublin Voivodeship
  - Lubelskie Centrum Diagnostyczne, Świdnik, Lublin Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw, Masovian Voivodeship
  - Bialystok - ClinicMed Daniluk, Nowak Spólka Jawna, Bialystok, Podlaskie Voivodeship
  - NZOZ Osteo Medic SC Artur Racewicz Jerzy Supronik, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Czestochowa - PRATIA - PPDS, Częstochowa, Silesian Voivodeship
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Medyczne Katowice - PRATIA - PPDS, Katowice
  - Centrum Medyczne Linden, Krakow
  - Krakowskie Centrum Medyczne, Krakow
  - MCM Krakow - PRATIA - PPDS, Krakow
  - Centrum Medyczne AMED, Warsaw
  - Centrum Medyczne Reuma Park NZOZ, Warsaw
  - Rheuma Medicus Specjalistyczne Centrum Reumatologii i Osteoporozy, Warsaw
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
- Serbia (4):
  - Institute of Rheumatology Belgrade - PPDS, Belgrade
  - Military Medical Academy, Belgrade
  - University Clinical Center of Serbia - PPDS, Belgrade
  - Clinical Centre of Vojvodina, Novi Sad

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 62 sites in 8 countries (Bulgaria, Estonia, Georgia, Hungary, Latvia, Poland, Serbia, and Mexico) screened at least one subject and 56 sites randomised at least one subject into the study.
Pre-assignment Details: The study included the Screening Period (28 days before randomization) that began after the participants had signed the written informed consent form. On Day 1 of the Main Treatment Period (MTP), subjects were randomly assigned in a 2:1:1 ratio to one of the 3 arms to receive one subcutaneous (SC) injection of European Union (EU) Prolia or MB09. Only those subjects who tolerated the initial 2 doses received the third dose and proceeded to the Transition/Safety Follow-up Period (TP).
Groups:
- MB09 (MTP): * Subjects randomised into MB09 group received one subcutaneous (SC) injection of MB09 (60 mg/mL) every 6 months (on Day 1, and Month 6).
  * MB09 (denosumab biosimilar): 60 mg/mL solution for injection in Prefilled Syringe (PFS).
  * Daily supplementation: at least 1000 mg elemental calcium and at least 400 IU of vitamin D.
- EU-Prolia (MTP): * Subjects randomised into Prolia-Prolia group received one SC injection of EU-Prolia® (60 mg/mL) every 6 months (on Day 1, and Month 6).
  * EU-Prolia®: 60 mg/mL solution for injection in PFS.
  * Daily supplementation: at least 1000 mg elemental calcium and at least 400 IU of vitamin D.
- MB09-MB09 (TP): * Subjects randomised into MB09-MB09 group received one subcutaneous (SC) injection of MB09 (60 mg/mL) every 6 months (on Day 1, Month 6, and Month 12).
  * MB09 (denosumab biosimilar): 60 mg/mL solution for injection in Prefilled Syringe (PFS).
  * Daily supplementation: at least 1000 mg elemental calcium and at least 400 IU of vitamin D.
- EU-Prolia-MB09 (TP): * Subjects randomised into Prolia-MB09 group received one SC injection of EU-Prolia® (60 mg/mL) every 6 months (on Day 1 and at Month 6) and one SC injection of MB09 at Month 12.
  * MB09 (denosumab biosimilar) and EU-Prolia®: 60 mg/mL solution for injection in PFS.
  * Daily supplementation: at least 1000 mg elemental calcium and at least 400 IU of vitamin D.
- EU Prolia-EU Prolia (TP): * Subjects randomised into Prolia-Prolia group received one SC injection of EU-Prolia® (60 mg/mL) every 6 months (on Day 1, Month 6 and Month12).
  * EU-Prolia®: 60 mg/mL solution for injection in PFS.
  * Daily supplementation: at least 1000 mg elemental calcium and at least 400 IU of vitamin D.
Period: Main Treatment Period (Day1 to Month 12)
Arm/Group | MB09 (MTP) | EU-Prolia (MTP) | MB09-MB09 (TP) | EU-Prolia-MB09 (TP) | EU Prolia-EU Prolia (TP)
Started (Note: Counts are presented according to treatment as randomised except for the safety analysis set (SAF), pharmacokinetics concentration Set (PKCS), and PK parameter Set (PKPS) where counts were presented according to the treatment received. One subject was not dosed per the randomisation schedule. This was handled as an intercurrent event.) | 281 | 277 | 0 | 0 | 0
Safety Analysis Set (SAF) | 277 | 278 | 0 | 0 | 0
Full Analysis Set (FAS) | 278 | 277 | 0 | 0 | 0
Modified Full Analysis Set (mFAS) | 258 | 266 | 0 | 0 | 0
Pharmacokinetics Parameter Set (PKPS) | 269 | 274 | 0 | 0 | 0
Pharmacokinetics Concentration Set (PKCS) | 277 | 278 | 0 | 0 | 0
Completed (Note that one subject randomly assigned to the MB09-MB09 arm did not receive the assigned treatment due to an isolated technical malfunction in the IRT system and instead received study treatment assigned to the Prolia Prolia arm throughout the study.) | 245 | 252 | 0 | 0 | 0
Not Completed | 36 | 25 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0
Not completed — unrelated medical conditions | 1 | 0 | 0 | 0 | 0
Not completed — subject dosed in error and did not meet eligibility criteria | 6 | 6 | 0 | 0 | 0
Not completed — other | 23 | 16 | 0 | 0 | 0
Period: Transition Period (M12 to M18)
Arm/Group | MB09 (MTP) | EU-Prolia (MTP) | MB09-MB09 (TP) | EU-Prolia-MB09 (TP) | EU Prolia-EU Prolia (TP)
Started (Note: Counts were presented according to treatment as randomised except for the SAF-TP, PKCS-TP, and PKPS-TP where counts were presented according to the treatment received. One subject was not dosed per the randomisation schedule. This was handled as an intercurrent event.) | 0 | 0 | 245 | 130 | 122
Safety Analysis Set for Transition Period (SAF-TP). | 0 | 0 | 244 | 130 | 123
Full Analysis Set for Transition Period (FAS-TP) | 0 | 0 | 245 | 130 | 122
Modified Full Analysis Set for Transition Period (mFAS-TP) | 0 | 0 | 233 | 127 | 121
Pharmacokinetic Concentration Set for Transition Period (PKCS-TP) | 0 | 0 | 244 | 130 | 123
Pharmacokinetic Parameter Set for Transition Period (PKPS-TP) | 0 | 0 | 228 | 126 | 111
Completed | 0 | 0 | 239 | 127 | 119
Not Completed | 0 | 0 | 6 | 3 | 3
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 3 | 2
Not completed — Burden of study procedures | 0 | 0 | 1 | 0 | 0
Not completed — Subject left the country | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAF) consisted of all randomised subjects who received at least one administration of study treatment.
Groups:
- MB09: •Subjects randomised into MB09 group received one subcutaneous (SC) injection of MB09 (60 mg/mL) every 6 months (on Day 1, and Month 6).
- EU-Prolia: •Subjects randomised into Prolia-Prolia group received one SC injection of EU-Prolia® (60 mg/mL) every 6 months (on Day 1, and Month 6).
- Total: Total of all reporting groups
Arm/Group | MB09 | EU-Prolia | Total
Number analyzed (Participants) | 277 | 278 | 555
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (6.00) | 65.9 (5.90) | 65.8 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 277 | 278 | 555
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race - White | 276 | 275 | 551
  Race - American Indian or Alaska Native | 1 | 3 | 4
  Ethnicity - Hispanic or Latino | 10 | 13 | 23
  Ethnicity - Not Hispanic or Latino | 267 | 265 | 532
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.62 (3.01) | 24.73 (3.06) | 24.68 (3.04)
Osteoporosis diagnosis duration [Mean (Standard Deviation); unit: years] | 2.6 (4.39) | 2.0 (3.89) | 2.3 (4.15)
Baseline BMD T-score at the lumbar spine [Count of Participants; unit: Participants] — The randomisation was stratified by baseline BMD T-score at the lumbar spine (≤ -3.0 and > -3.0 SD, with the worst prognosis bellow or equal to - 3 (≤ -3.0) and the better prognosis higher than -3 (> -3.0).
  Participants
    > -3.0 group | 144 | 143 | 287
    ≤ -3.0 group | 133 | 135 | 268
Lumbar spine BMD [Mean (Standard Deviation); unit: g/cm^2] | 0.766 (0.0878) | 0.773 (0.0862) | 0.770 (0.0870)
Total hip BMD [Mean (Standard Deviation); unit: g/cm^2] | 0.731 (0.0973) | 0.745 (0.0946) | 0.738 (0.0961)
Femur neck BMD [Mean (Standard Deviation); unit: g/cm^2] | 0.672 (0.1085) | 0.685 (0.1084) | 0.679 (0.1086)
Prior use of bisphosphonates [Count of Participants; unit: Participants]
  Yes | 25 | 21 | 46
  No | 252 | 257 | 509
Previous Fractures in the Medical History [Count of Participants; unit: Participants]
  Yes | 108 | 102 | 210
  No | 169 | 176 | 345
Menopause duration [Mean (Standard Deviation); unit: years] | 16.4 (7.05) | 16.9 (7.35) | 16.7 (7.20)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Percentage Change From Baseline (%CfB) in Lumbar Spine Bone Mineral Density (LS-BMD) at 52 Weeks - Modified Full Analysis Set (mFAS)
Description: To demonstrate equivalent efficacy of MB09 to EU Prolia in postmenopausal women with osteoporosis in terms of lumbar spine BMD at Week 52 (Month 12). The main analysis method was on the mFAS using a mixed model for repeated measures (MMRM) fitted to the composite %CfB lumbar spine BMD at Month 6 and Month 12, without any imputation of missing data. Bone mineral density was assessed by dual-energy X-ray absorptiometry (DXA) and assessments of the lumbar spine (L1 to L4) were performed at a central imaging vendor.
Time Frame: Baseline (Screening), up to Week 52
Population: Modified Full Analysis Set (mFAS) is a subset of subjects in the FAS who met all eligibility criteria. The mFAS term defined a set at the data point level which included a data record at each timepoint for all eligible subjects in the FAS but excluded data observed after the first occurrence of those intercurrent events (ICEs) where a hypothetical strategy was taken (eg, missing a dose, errors or deviations in dosing, or receipt of any prohibited therapies or other osteoporosis medication).
Measure: Least Squares Mean (Standard Error); unit: Percentage change (%)
Groups:
- MB09: A total of 2 subcutaneous administration of 60 mg MB09 (proposed denosumab biosimilar) on Day 1 and Month 6 in the Main Treatment Period (MTP).
- EU-Prolia: A total of 2 subcutaneous administration of 60 mg Prolia on Day 1 and Month 6 in the Main Treatment Period (MTP).
Arm/Group | MB09 | EU-Prolia
Number analyzed (Participants) | 233 | 250
Percentage change (%) | 5.86 (0.26) | 5.66 (0.25)
Statistical Analysis 1: Comparison: MB09 vs EU-Prolia; Test type: Equivalence — The estimated mean difference in %CfB lumbar spine BMD at Month 12 was presented with 95% CI and equivalence was concluded if this fell within the predefined equivalence margin of [-1.45%, 1.45%]; Mixed Models Analysis — Mixed-model for repeated measures (MMRM); MMRM included treatment, with stratification variables as classification factors and baseline BMD as a continuous covariate; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.51 to 0.91]

2. Secondary Outcome: Efficacy: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (LS-BMD) at Week 52 - Full Analysis Set (FAS)
Description: Difference in means (MB09-Prolia) in the %CfB in lumbar spine BMD after 12 months in postmenopausal women with osteoporosis treated with SC denosumab injections every 6 months. This included all subjects and data records irrespective of failed eligibility criteria, receipt of prohibited medications, discontinued treatment for any reason, had errors or deviations in dosing, or receipt of both doses. Estimation was via Multiple Imputation (MI) and ANCOVA on the FAS. Since the retrieved dropout rate was low, a treatment-failure (TF) penalty was applied to the imputed values at Month 12 for those subjects who received only one dose of the study treatment to centre the distribution of each subject's %CfB values around their baseline level. Bone density measurements were performed by DXA. All DXA scans were submitted to a central imaging vendor for analysis.
Time Frame: Baseline (screening), up to Week 52
Population: The Full Analysis Set (FAS) consisted of all consenting randomised subjects who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Percentage change (%)
Arm/Group | MB09 | EU-Prolia
Number analyzed (Participants) | 278 | 277
Percentage change (%) | 5.40 (0.26) | 5.38 (0.26)
Statistical Analysis 1: Comparison: MB09 vs EU-Prolia; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; ANCOVA included terms for treatment, with stratification variables as classification factors and baseline BMD included as a continuous covariate; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.69 to 0.74] — The estimated mean difference in %CfB lumbar spine BMD results was pooled using Rubin's methods and presented with 95% CI

3. Secondary Outcome: Efficacy: Percentage Change From Baseline (%CfB) in Lumbar Spine at Month 6 and Total Hip and Femur Neck BMD at Month 6 and Month12 - MMRM on mFAS
Description: To assess the efficacy of MB09 to EU-Prolia in postmenopausal women with osteoporosis in terms of Lumbar Spine at Month 6 and Total Hip and Femur Neck BMD at Month 6 and Month12. The difference in means in %CfB in lumbar spine BMD between MB09 and Prolia at Month 6 and Total Hip and Femur Neck at Month 6 and Month 12 from an MMRM presented for the mFAS. Bone density measurements were performed by DXA. All DXA scans were submitted to a central imaging vendor for analysis.
Time Frame: Baseline (screening), Month 6 and Month 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage change (%)
Groups:
- MB09: Subcutaneous administration of 60 mg MB09 (proposed denosumab biosimilar) every 6 months, on Day 1 and Month 6 in the Main Treatment Period (MTP).
- EU-Prolia: Subcutaneous administration of 60 mg Prolia every 6 months, on Day 1 and Month 6 in the Main Treatment Period (MTP).
Arm/Group | MB09 | EU-Prolia
Number analyzed (Participants) | 258 | 266
percentage change (%)
  Total Hip - Month 12: number analyzed (Participants) | 232 | 252
  Total Hip - Month 12 | 3.37 (0.18) | 3.28 (0.17)
  Femur Neck - Month 12: number analyzed (Participants) | 232 | 252
  Femur Neck - Month 12 | 2.75 (0.23) | 2.39 (0.23)
  Lumbar Spine - Month 6: number analyzed (Participants) | 246 | 258
  Lumbar Spine - Month 6 | 4.03 (0.23) | 3.96 (0.22)
  Total Hip - Month 6: number analyzed (Participants) | 241 | 257
  Total Hip - Month 6 | 2.29 (0.16) | 2.46 (0.16)
  Femur Neck - Month 6: number analyzed (Participants) | 241 | 257
  Femur Neck - Month 6 | 2.18 (0.22) | 1.93 (0.21)

4. Secondary Outcome: Efficacy: Percentage Change From Baseline (%CfB) in Lumbar Spine BMD at Month 6 and Total Hip and Femur Neck BMD at Month 6 and 12 - ANCOVA on FAS
Description: To assess the efficacy of MB09 to EU-Prolia in postmenopausal women with osteoporosis in terms of the difference in means (MB09-Prolia) in the %CfB in Lumbar Spine BMD at Month 6 and Total Hip and Femur Neck BMD at Month 6 and 12 in postmenopausal women with osteoporosis treated with SC denosumab injections every 6 months. This included all subjects and data records irrespective of failed eligibility criteria, receipt of prohibited medications, discontinued treatment for any reason, had errors or deviations in dosing, or receipt of both doses. Bone density measurement were performed by DXA. All DXA scans were submitted to a central imaging vendor for analysis.
Time Frame: Baseline (screening), Month 6, Month 12.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change (%)
Arm/Group | MB09 | EU-Prolia
Number analyzed (Participants) | 278 | 277
percentage change (%)
  Total Hip - Month 12: number analyzed (Participants) | 254 | 260
  Total Hip - Month 12 | 3.31 (0.17) | 3.27 (0.17)
  Femur Neck- Month 12: number analyzed (Participants) | 254 | 260
  Femur Neck- Month 12 | 2.70 (0.23) | 2.38 (0.22)
  Lumbar Spine - Month 6 | 3.82 (0.22) | 3.92 (0.22)
  Total Hip - Month 6: number analyzed (Participants) | 262 | 270
  Total Hip - Month 6 | 2.28 (0.16) | 2.49 (0.16)
  Femur Neck - Month 6: number analyzed (Participants) | 262 | 270
  Femur Neck - Month 6 | 2.18 (0.21) | 1.92 (0.21)

5. Secondary Outcome: Pharmacodynamics: Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen (sCTX) Area Under the Effect Curve From Zero to 6 Months (AUEC0-6 Months) After First Dose - Modified Full Analysis Set (mFAS)
Description: Geometric meant (geometric CV%) sCTX Area under the effect curve from zero to 6 months (AUEC0-6 months) after first dose in postmenopausal women with osteoporosis treated with SC denosumab injections every 6 months assuming all women received their first denosumab dose without any errors in dosing and without receipt of any prohibited therapies or other osteoporosis medications up to 6 months after first dose.
Time Frame: Baseline (pre-dose Day 1), up to Month 6.
Population: Modified Full Analysis Set (mFAS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*pg/mL
Arm/Group | MB09 | EU-Prolia
Number analyzed (Participants) | 218 | 228
day*pg/mL | 12300 (49.7) | 12400 (44.1)
Statistical Analysis 1: Comparison: MB09 vs EU-Prolia; Test type: Equivalence — Equivalence criteria (analysis set mFAS): 95% CI for ratio of geometric LS mean ratios contained in acceptance limits (80.00%, 125.00%); ANCOVA; ANCOVA model including log-transformed baseline sCTX as a continuous covariate with treatment and stratification variables as fixed effects; Ratio of Geometric means = 99.91, 95% CI 2-sided [91.99 to 108.52]

6. Secondary Outcome: Pharmacodynamics: %CfB Area Under the Percent Inhibition Curve From Time Zero to 6 Months (AUIC0-6 Months) in sCTX - on mFAS
Description: AUIC0-6 months = Area under the inhibition curve for % change from baseline sCTX concentrations from time zero to 6 months
Time Frame: Baseline (pre-dose Day 1), up to Month 6.
Population: Modified Full Analysis Set (mFAS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day* %
Arm/Group | MB09 | EU-Prolia
Number analyzed (Participants) | 218 | 228
day* % | 15100 (17.4) | 15300 (13.6)
Statistical Analysis 1: Comparison: MB09 vs EU-Prolia; Test type: Equivalence — Biosimilarity with respect to PD was concluded if the 95% CI for the test (MB09) to reference (EU-Prolia) ratios of the geometric LS means was contained within the [80.00%, 125.00%] interval; ANCOVA; Ratio of Geometric means = 99.13, 95% CI 2-sided [96.31 to 102.02]

7. Secondary Outcome: Pharmacokinetics: Maximum Observed Serum Concentration (Cmax) of Denosumab After First Dose Study Treatment (Pharmacokinetic Parameter Analysis Set)
Description: To assess the PK profile of MB09 compared with EU-Prolia following the first dose, maximum Observed Serum Concentration (Cmax) of Denosumab After First Dose study treatment (Pharmacokinetic Parameter Analysis Set).
Time Frame: Baseline (pre-dose Day 1), up to Month 6
Population: Pharmacokinetic Parameter Analysis Set (PKPS) comprises all subjects who have at least three measurable concentrations in PKCS which must include Day 11 to allow for reliable estimation of both Cmax and AUC0-6 months.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MB09 | EU-Prolia
Number analyzed (Participants) | 269 | 273
ng/mL | 5960 (31.1) | 5700 (35.9)
Statistical Analysis 1: Comparison: MB09 vs EU-Prolia; Test type: Equivalence — Equivalence criteria (on Pharmacokinetic Parameter Analysis Set): the 95% CIs around the geometric LS mean contained in the acceptance limits (80.00%, 125.00%); ANCOVA; Cmax was analysed on the log scale by ANCOVA. The model included treatment and stratification variables as fixed effects; LS Geometric Mean Ratio = 104.13, 95% CI 2-sided [98.83 to 109.71]

8. Secondary Outcome: Pharmacokinetics: To Assess the PK Profile of MB09 Compared With EU Prolia (AUC0-6 Months) Following the First Dose
Description: Area under the concentration-time curve from time zero to 6 months analysed on the log scale by ANCOVA. The model will include treatment and stratification variables (baseline BMD T-score at the lumbar spine (≤ -3.0 and > -3.0 SD), body mass index (< 25 and ≥ 25 kg/m2), age at study entry (≥ 55 to < 68 years versus ≥ 68 to ≤ 80 years) and prior bisphosphonate medication use at study entry (prior use of bisphosphonates versus no prior bisphosphonate use as fixed effects. The estimated mean difference with 95% CI will be back-transformed to give the ratio of geometric means (MB09/EU-Prolia) with 95% CI following the first dose in the Main Treatment Period.
Time Frame: Baseline (pre-dose Day 1), up to Month 6.
Population: Pharmacokinetic Parameter Analysis Set (PKPS) comprises all subjects who have at least three measurable concentrations in PKCS wich must include Day 11 to allow for reliable estimation of both Cmax and AUC0-6 months.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | MB09 | EU-Prolia
Number analyzed (Participants) | 256 | 260
day*ng/mL | 360,000 (36.5) | 337000 (39.5)
Statistical Analysis 1: Comparison: MB09 vs EU-Prolia; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; ANCOVA; AUC0-6 months was analysed on the log scale by ANCOVA. The model included treatment and stratification variables as fixed effects; LS Geometric Mean Ratio = 106.06, 95% CI 2-sided [99.84 to 112.66]

9. Secondary Outcome: Safety: Overall Summary of Adverse Events - Main Treatment Period - Safety Analysis Set (SAF) and Safety Analysis Set for Transition Period (SAF-TP)
Description: For Main Treatment Period, treatment-emergent adverse event (TEAE) was an event observed after first dose on Day 1 until Month 12 and no more than 6 months after the last dose in case of early treatment discontinuation unless the TEAE was considered as related to the study treatment by investigator. For Transition Period, TEAE was an event observed after the third dose of study treatment at Month 12 until Month 18. Throughout the study, TEAE was an event observed after first dose on Day 1 until Month 18.
Time Frame: From first administration of study treatment on Day 1 until Month 18
Population: The Safety Analysis Set (SAF) and Safety Analysis Set for Transition Period (SAF-TP)
Measure: Count of Participants; unit: Participants
Groups:
- Main Treatment Period: MB09: From first administration of study treatment on Day 1 until Month 12 (pre-dose) displayed for MB09 group.
- Main Treatment Period: EU-Prolia: From first administration of study treatment on Day 1 until Month 12 (pre-dose) displayed for EU-Prolia group.
- Throughout the Study: MB09-MB09: Cumulative safety data throughout the study (baseline to the end of Transition Period [Month 18]) displayed for MB09-MB09 group.
- Throughout the Study: Prolia-MB09: Cumulative safety data throughout the study (baseline to the end of Transition Period [Month 18]) displayed for Prolia-MB09 group.
- Throughout the Study: Prolia-Prolia: Cumulative safety data throughout the study (baseline to the end of Transition Period [Month 18]) displayed for Prolia-Prolia group.
Arm/Group | Main Treatment Period: MB09 | Main Treatment Period: EU-Prolia | Throughout the Study: MB09-MB09 | Throughout the Study: Prolia-MB09 | Throughout the Study: Prolia-Prolia
Number analyzed (Participants) | 277 | 278 | 277 | 140 | 138
Participants
  Any TEAEs | 161 | 150 | 180 | 87 | 75
  Any study treatment-related TEAEs | 41 | 24 | 45 | 11 | 17
  Any serious TEAEs | 19 | 13 | 21 | 11 | 4
  Any study treatment-related serious TEAEs | 1 | 1 | 1 | 0 | 1

10. Secondary Outcome: Safety: New Clinical Bone Fractures - TEAEs (Throughout the Study - From Day 1 Untill Month 18)
Description: For the Main Treatment Period, TEAE was an event observed after first dose on Day 1 until Month 12 and no more than 6 months after the last dose in case of early treatment discontinuation unless the TEAE was considered as related to the study treatment by investigator. For Transition Period, TEAE was an event observed after the third dose of study treatment at Month 12 until Month 18. Throughout the study, TEAE was an event observed after first dose on Day 1 until Month 18.
Time Frame: All participants in the Main Treatment Period and Transition Period (From Day 1 untill Month 18)
Population: Safety Analysis Set (SAF) and Safety Analysis Set for Transition Period (SAF-TP)
Measure: Count of Participants; unit: Participants
Groups:
- Throughout the Study: EU Prolia-MB09: Cumulative safety data throughout the study (baseline to the end of Transition Period [Month 18]) displayed for EU Prolia-MB09 group.
- Throughout the Study: EU Prolia- EU Prolia: Cumulative safety data throughout the study (baseline to the end of Transition Period [Month 18]) displayed for EU Prolia- EU Prolia group.
Arm/Group | Throughout the Study: MB09-MB09 | Throughout the Study: EU Prolia-MB09 | Throughout the Study: EU Prolia- EU Prolia
Number analyzed (Participants) | 277 | 140 | 138
Participants
  Number of subjects with at least one fracture TEAE (any bone) | 12 | 6 | 4
  Number of subjects with at least one Vertebral fracture | 3 | 2 | 1
  Number of subjects with at least one Hip fracture | 1 | 1 | 0
  Number of subjects with at least one Pelvic fracture | 1 | 0 | 0

11. Secondary Outcome: Overall Incidence of Antidrug Antibodies (ADA) - Safety Analysis Set (SAF) and Safety Analysis Set for Transition Period (SAF-TP)
Description: Number of subjects experiencing treatment-induced immunogenicity: Binding and neutralising serum denosumab antibodies from baseline up to and including Month 18. Analysis of immunogenicity data will be based on ADA evaluable subjects defined as all SAF or SAF-TP subjects with baseline and at least one post-baseline immunogenicity assessment within the Main Treatment Period or the Transition Period. The formation of ADAs against MB09 or EU-Prolia was assessed in blood samples.
Time Frame: From baseline (pre-dose) up to and including Month 18.
Population: Safety Analysis Set (SAF) and Safety Analysis Set for Transition Period (SAF-TP)
Measure: Count of Participants; unit: Participants
Arm/Group | Throughout the Study: MB09-MB09 | Throughout the Study: EU Prolia-MB09 | Throughout the Study: EU Prolia- EU Prolia
Number analyzed (Participants) | 277 | 140 | 138
Participants
  ADA positive | 1 | 3 | 3
  NAb positive | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Subject incidence of TEAEs up to and including Month 18.
Description: For Main Treatment Period, TEAE was an event observed after first dose on Day 1 until Month 12 and no more than 6 months after the last dose in case of early treatment discontinuation unless the TEAE was considered as related to the study treatment by investigator. For Transition Period, TEAE was an event observed after the third dose of study treatment at Month 12 until Month 18. Throughout the study, TEAE was an event observed after first dose on Day 1 until Month 18.
Groups:
- Throughout the Study: EU Prolia-EU Prolia: Cumulative safety data throughout the study (baseline to the end of Transition Period [Month 18]) displayed for EU Prolia-EU Prolia group.
Arm/Group | Main Treatment Period: MB09 | Main Treatment Period: EU-Prolia | Throughout the Study: MB09-MB09 | Throughout the Study: EU Prolia-MB09 | Throughout the Study: EU Prolia-EU Prolia
All-Cause Mortality (participants affected / at risk) | 0/277 | 0/278 | 1/277 | 0/140 | 0/138
Serious Adverse Events (participants affected / at risk) | 19/277 | 13/278 | 21/277 | 11/140 | 4/138
Other Adverse Events (participants affected / at risk) | 120/277 | 120/278 | 180/277 | 87/140 | 75/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Treatment Period: MB09 (N=277) | Main Treatment Period: EU-Prolia (N=278) | Throughout the Study: MB09-MB09 (N=277) | Throughout the Study: EU Prolia-MB09 (N=140) | Throughout the Study: EU Prolia-EU Prolia (N=138)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Toxic goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Treatment Period: MB09 (N=277) | Main Treatment Period: EU-Prolia (N=278) | Throughout the Study: MB09-MB09 (N=277) | Throughout the Study: EU Prolia-MB09 (N=140) | Throughout the Study: EU Prolia-EU Prolia (N=138)
Upper respiratory tract infection (Infections and infestations) | 20 (20) | 20 (22) | 25 (30) | 13 (15) | 12 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (16) | 15 (15) | 17 (18) | 5 (6) | 10 (10)
COVID-19 (Infections and infestations) | 14 (14) | 15 (15) | 21 (21) | 11 (11) | 10 (10)
Blood parathyroid hormone increased (Investigations) | 11 (12) | 4 (4) | 11 (12) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 10 (10) | 6 (6) | 10 (10) | 4 (4) | 6 (6)
Nasopharyngitis (Infections and infestations) | 10 (10) | 23 (23) | 15 (15) | 15 (16) | 11 (11)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (12) | 10 (13) | 11 (14) | 4 (5) | 7 (9)
Urinary tract infection (Infections and infestations) | 9 (13) | 9 (12) | 18 (23) | 8 (12) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 4 (4) | 8 (8) | 2 (2) | 3 (3)
Hypothyroidism (Endocrine disorders) | 6 (6) | 6 (6) | 7 (8) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (7) | 7 (8) | 5 (5) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 6 (6) | 5 (6) | 8 (8) | 4 (5) | 3 (3)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 7 (9) | 3 (4) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 7 (8) | 3 (3) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (7) | 5 (5) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (8) | 2 (2) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 2 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 4 (4)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (5)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT05338086/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT05338086/SAP_001.pdf